CLINICAL TRIAL: NCT02646761
Title: interACTION: A Portable Joint Function Monitoring and Training System for Remote Rehabilitation Following Total Knee Arthroplasty
Brief Title: interACTION: A Portable Joint Function Monitoring and Training System for Remote Rehabilitation Following TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Irrgang (Other)
Responsible Party: Sponsor-Investigator, James J. Irrgang, PhD, PT, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO15060281
Record Dates: First submitted 2015-08-14; First posted 2016-01-06 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation with InterACTION (Experimental): After total knee arthroplasty, subjects will undergo physical therapy 1 time per week supplemented by home exercise program with InterACTION device.
  Interventions: Device: InterACTION
- Standard Physical Therapy (Other): After total knee arthroplasty, subjects will undergo standard of care physical therapy 2 times per week with standard home exercise program.
  Interventions: Other: Standard of Care Physical Therapy

INTERVENTIONS:
Device: InterACTION — InterACTION guided home exercise program paired with standard of care physical therapy
  Arms: Rehabilitation with InterACTION
Other: Standard of Care Physical Therapy — Physical therapy rehabilitation program
  Arms: Standard Physical Therapy

SUMMARY:
The purpose of this study is to determine if home-based therapy with monitoring via telemedicine can overcome many barriers to compliance and improve rehabilitation. Patients undergoing total knee arthroplasty will be followed for 10 weeks during their outpatient physical therapy course. Subjects will undergo standard physical therapy or physical therapy paired with InterACTION for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 40 to 80 years of age;
2. Have undergone primary unilateral total knee arthroplasty;
3. Being referred for post-operative outpatient physical therapy;
4. Agree to and able to perform pre-defined exercises that they would normally perform in a physical rehabilitation program.

Exclusion Criteria:

1. Patients with BMI >40 at the time of surgery;
2. Individuals who are not free of any other co-disability or comorbidity that would specifically impede disallow or otherwise hinder performance of rehabilitation exercises;
3. Individuals who cannot physically receive or understand audio and visual feedback from the joint motion tracking system during or after performance of rehabilitation exercises;
4. Individuals who are discharged post-operatively to a skilled nursing facility instead of to their residence;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Bell KM, Onyeukwu C, Smith CN, Oh A, Devito Dabbs A, Piva SR, Popchak AJ, Lynch AD, Irrgang JJ, McClincy MP. A Portable System for Remote Rehabilitation Following a Total Knee Replacement: A Pilot Randomized Controlled Clinical Study. Sensors (Basel). 2020 Oct 27;20(21):6118. doi: 10.3390/s20216118. PMID 33121204

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 subjects were assessed for eligibility for the study. Nine were deemed ineligible and 38 were randomized into one of the 2 study arms. Subjects were recruited and randomized prior to surgery & the baseline assessment was done approximately 2 to 4 weeks after surgery.
Groups:
- Rehabilitation With InterACTION: Subjects underwent a rehabilitation program with InterACTION.
- Standard Physical Therapy: Subjects underwent standard of care physical therapy.
Period: Overall Study
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Started | 18 | 20
Subject Withdrew Before Baseline | 5 | 8
Baseline Assessment | 13 | 12
5-week Assessment | 12 | 10
Completed | 10 | 10
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Population: Baseline assessments were performed approximately 2 to 4 weeks after subjects underwent TKA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (6.6) | 65.9 (7.6) | 65.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Marital status [Count of Participants; unit: Participants]
  Married | 11 | 8 | 19
  Separated | 0 | 1 | 1
  Single | 2 | 1 | 3
  Widowed | 0 | 2 | 2
Education [Count of Participants; unit: Participants]
  Some high school | 0 | 0 | 0
  High school grad | 2 | 3 | 5
  Some college | 0 | 4 | 4
  College graduate | 4 | 2 | 6
  Some graduate school | 1 | 2 | 3
  Graduate degree | 6 | 1 | 7
Employment Status [Count of Participants; unit: Participants]
  Retired due to health | 1 | 0 | 1
  Retired not due to health | 7 | 6 | 13
  Temporary retired due to health | 1 | 1 | 2
  Semi-retired | 1 | 0 | 1
  Regular full time | 3 | 4 | 7
  Regular part time | 0 | 1 | 1
Current Smoker [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Value Was Evaluated as the Ratio of Change in the Activities of Daily Living Scale Score to the Costs of Rehabilitation.
Description: The value was calculated the ratio of the difference between the 10 week and baseline Activities of Daily Living Scale (ADLS) of the Knee Outcome Survey divided by the total charges for the physical therapy treatment sessions. The ADLS is a 14-item measure of symptoms and activity limitations for individuals with a variety of knee impairments. Items are scored from 0 to 4, and the total score is the sum of all the items divided by 70 and multiplied by 100. The ADLS score ranges from 0 to 100 with higher scores representing less symptoms and greater levels of activity. Higher ratio of the change in the ADLS score to the costs for rehabilitation represents greater value.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Number analyzed (Participants) | 10 | 10
ratio | 0.013 (0.007) | 0.018 (0.009)

2. Secondary Outcome: Number of Participants That Complied With Rehabilitation Program
Description: Compliance with the use of the InterACTION device was measured by reports generated from the device. Subjects in the Standard Physical Therapy Group completed exercise logs that were monitored at each study visit.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Number analyzed (Participants) | 10 | 10
Participants
  Greater than 90% | 6 | 5
  71-90% | 4 | 2
  51-70% | 0 | 0
  31-50% | 0 | 1
  0-30% | 0 | 0
  Missing Compliance Data | 0 | 2

3. Secondary Outcome: Number of Subjects Satisfied With InterACTION Device
Description: Subjects in the interACTION group were asked "Would you consider using the InterACTION device if you had to do rehabilitation again in the future?"
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation With InterACTION
Number analyzed (Participants) | 11
Participants
  Yes | 11
  No | 0

4. Secondary Outcome: Performance Based Outcome Measures
Description: The performance based measures included the 6-minute walk test (measured as distance in meters); stair climb test (measured as time in seconds divided by the number of steps); timed up and go test (measured in seconds); and unilateral balance test (measured in seconds). To combine the 4 performance-based outcome measures into a single composite score, the score for each test was converted to a z score (individual's score - overall mean)/overall standard deviation. As such, the z-score represents the number of SD deviations an individual's score is above or below the overall study mean. A z-score of 0 implies the participants score is the same as the mean score. A z-score of 0.1 would indicate that the participant's z score is .1 (10%) of a standard deviation above or below the overall mean. The average of the z scores for each performance-based outcome measure as the unit of analysis.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Number analyzed (Participants) | 10 | 10
z-score | -0.0071 (1.02) | 0.028 (0.64)

5. Secondary Outcome: Range of Motion (Extension)
Description: Extension of both knees was measured with a goniometer and the side-to-side difference was expressed in degrees.
Time Frame: baseline and 10 weeks
Population: The total number analyzed represents the subjects that did not drop out of the study and completed the 10 weeks follow-up assessment.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Number analyzed (Participants) | 10 | 10
degrees
  Baseline Active Extension | 5.3 (5.6) | 1.1 (3.4)
  10 weeks Active Extension | 1.6 (2.5) | 1.7 (2.5)

6. Secondary Outcome: Range of Motion (Flexion)
Description: Flexion of both knees was measured with a goniometer and the side-to-side difference was expressed in degrees.
Time Frame: baseline and 10 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
Number analyzed (Participants) | 10 | 10
degrees
  Baseline Active Flexion | 93.0 (17.6) | 91.5 (19.3)
  10 weeks Active Flexion | 120.8 (8.6) | 123.1 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of the intervention until 10 weeks follow-up.
Arm/Group | Rehabilitation With InterACTION | Standard Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT02646761/Prot_SAP_000.pdf